CLINICAL TRIAL: NCT06879314
Title: Investigation of Motor Development and Sensory Processing Skills in Children Diagnosed With Congenital Muscular Torticollis
Brief Title: Development in Children Diagnosed With Congenital Muscular Torticollis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Gazi University
Other Study IDs: torticollis RZ
Record Dates: First submitted 2025-03-10; First posted 2025-03-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-03

CONDITIONS: Torticollis Congenital; Motor Development; Sensory Integration Dysfunction
Keywords: Torticollis; motor development; sensory processing skills; infant
MeSH Terms: conditions — Congenital torticollis; Torticollis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- torticollis: Twenty children with congenital muscular torticollis diagnosis, between 0-12 months of age, with parental consent, without any vision or hearing problems, will be included in the study.
- Healthy infants: A control group of 20 healthy children without congenital muscular torticollis will be formed.

SUMMARY:
It has been thought that head position may affect the shoulder, rib cage and abdominal muscles, which may have a negative effect on posture control and movement development, sensory-motor coordination and cause retardation in gross motor function. For these reasons, children with congenital muscular torticollis should be evaluated comprehensively in the early period. This study, which was planned to evaluate the motor development and sensory processing of children with torticollis, was designed according to the lack of literature.

DETAILED DESCRIPTION:
Congenital muscular torticollis (CMT) is a common postural deformity that occurs shortly after birth and is typically characterized by ipsilateral cervical lateral flexion and contralateral cervical rotation due to unilateral shortening of the sternocleidomastoid (SCM) muscle. It is a non-neurological postural disorder that usually affects 3% to 16% of infants. Theories such as intrauterine stenosis, vascular causes, fibrosis of the peripartum hemorrhage area, difficult labor, and primary myopathy of the SCM muscle have been put forward for its causes. In tissue samples taken after surgery, edema, degeneration of muscle fibers, and fibrosis have been reported. It is thought that CMT affects the muscles as well as head and facial development, causing various asymmetries, delays in gross motor functions, and disorders in posture and balance control. A bent neck position can cause plagiocephaly. Characteristic craniofacial deformities include asymmetry in the brow and cheekbones, deviation of the chin and nose tip, inferior orbital abnormality on the affected side, asymmetry in ear placement, and shortening of the vertical dimension of the ipsilateral face. In later periods, it has been shown that it may cause asymmetry in the use of the upper extremities, delay in gross motor functions, and effects on posture and balance control in children. It is thought that head position may affect the shoulder, rib cage, and abdominal muscles, which may have a negative effect on posture control and movement development, sensory-motor coordination, and cause gross motor function retardation. For these reasons, children with congenital muscular torticollis should be evaluated comprehensively in the early period. This study, which was planned to evaluate the motor development and sensory processing of children with CMT, was designed according to the lack of literature.

ELIGIBILITY:
Inclusion Criteria:

* Infants diagnosed with congenital torticollis between 0-12 months of age,
* with parental consent,

Exclusion Criteria:

* Children with chromosomal abnormalities,
* serious congenital problems,
* vision-hearing problem
* children whose parents do not volunteer for the study will not be included in the study.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Congenital muscular torticollis (CMT) is a common postural deformity that appears shortly after birth and is typically characterized by ipsilateral cervical lateral flexion and contralateral cervical rotation due to unilateral shortening of the sternocleidomastoid (SCM) muscle. It is a non-neurological postural disorder that usually affects 3% to 16% of infants. CMT is the third most common musculoskeletal disorder of infancy, affecting 3.9% to 16% of infants. It develops due to unilateral shortening of the SCM, regardless of whether there is a mass in the SCM. CMT is characterized by lateral flexion of the affected SCM to the ipsilateral side and rotation to the contralateral side.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scale | Second Edition | 1-12 months
  It is planned to use Peabody Motor Development Scale-2 to evaluate motor development. The test is designed to determine developmental delays in children between 0-72 months. It is used to evaluate the motor development of children with separate tests and rating scales for both gross motor skills and fine motor skills. Six subtests, reflexes, Stationary, Locomotion, Object Manipulation, Grasping, and Visual-Motor Integration, collectively measure a broad spectrum of motor functions including postural control, locomotor abilities, object manipulation, and hand-eye coordination. The subtests generate three composite scores: the Gross Motor Quotient, Fine Motor Quotient, and Total Motor Quotient, offering a comprehensive evaluation of a child's motor competence. Notably, higher scores on the Peabody Motor Development Scale-2 reflect superior motor performance, indicating better developmental outcomes.
Test of Sensory Functions in Infants | 1-12 months
  It was planned to use the Test of Sensory Functions in Infants to evaluate the sensory development of infants. Test of Sensory Functions in Infants is frequently used to evaluate the sensory processing functions of infants aged 4-18 months. It is used to determine whether an infant has a sensory processing problem and to what extent. It consists of 24 items.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia ZORLULAR, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeGangi, G.A. and S.I. Greenspan, Test of sensory functions in infants (TSFI). 1989: Western Psychological Services Los Angeles
- [Background] Folio, M.R. and R.R. Fewell, Peabody developmental motor scales and activity cards. 1983: DLM Teaching
- [Background] Ohman A, Nilsson S, Lagerkvist AL, Beckung E. Are infants with torticollis at risk of a delay in early motor milestones compared with a control group of healthy infants? Dev Med Child Neurol. 2009 Jul;51(7):545-50. doi: 10.1111/j.1469-8749.2008.03195.x. Epub 2009 Jan 26. PMID 19191832
- [Derived] Zorlular R, Burak SE, Beyoglu R, Elbasan B. Motor development and sensory processing skills in infants with congenital muscular torticollis: a cross-sectional study. Eur J Pediatr. 2025 Sep 23;184(10):630. doi: 10.1007/s00431-025-06457-2. PMID 40986093